CLINICAL TRIAL: NCT02472041
Title: Effectiveness of Reanimator Muller in Patients With Chest Tube
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Ana Paula Ragonete dos Anjos, principal investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20300313.9.0000.5404
Record Dates: First submitted 2015-05-21; First posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Mechanical Ventilation Complication
Keywords: chest drain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reanimator Group (Experimental): Reanimator of Muller Group (intermittent positive pressure): Patients allocated to this group received intermittent positive pressure breathing (resuscitator Muller, Engemed, Brazil), adjusting the positive pressure around 1.5 kgf / cm2, which corresponds to 15 20 cm / H2O, positive pressure was applied through a face mask (Respironics®), which was connected in a circuit extending along the Muller Resuscitator equipment applied continuously for four series 10 of the patient breaths active and with an interval of two minutes between them in Fowler 45 position
  Interventions: Device: Reanimator group
- Control Group (Experimental): Control Group: In position Fowler 45, patients assigned to this group was administered as treatment lung expansion exercises using the incentive inspiratory flow (Respiron, NCS, Mexico) and concomitantly blocking contralateral to the drain maneuvers were performed, compression / decompression associated with the incentive spirometry (Respiron) consisting of 4 sets of 10 active patient breaths with an interval of two minutes between sets. Since the load of the respiratory stimulator will be zero throughout treatment (Table 1). Guidelines to the active, progressive and early mobilization.
  Interventions: Device: Control

INTERVENTIONS:
Device: Reanimator group — Resuscitator of Muller Group (intermittent positive pressure): Patients allocated to this group received intermittent positive pressure breathing (resuscitator Muller, Engemed, Brazil), adjusting the positive pressure around 1.5 kgf / cm2, which corresponds to 15 20 cm / H2O, positive pressure was applied through a face mask (Respironics®).
  Arms: Reanimator Group
Device: Control — Control Group: In position Fowler 45, patients assigned to this group was administered as treatment lung expansion exercises using the incentive inspiratory flow (Respiron, NCS, Mexico) and concomitantly blocking contralateral to the drain maneuvers were performed, compression / decompression associated with the incentive spirometry (Respiron) consisting of 4 sets of 10 active patient breaths with an interval of two minutes between sets. Since the load of the respiratory stimulator will be zero throughout treatment. Guidelines to the active, progressive and early mobilization.
  Arms: Control Group

SUMMARY:
This study evaluates the comparison of two of re-expansion pulmonary physiotherapy in patients with chest tube. The study group received intermittent positive pressure intervention and the control group received incentive spirometry intervention associated with manual operation.

DETAILED DESCRIPTION:
All the re-expansion methods increase lung volume increasing gradient of transpulmonary pressure (PL) representing the difference alveolar pressure and pleural pressure. Spontaneous deep breath increases the PL by reducing pleural pressure (active breathing exercises, breathing supporters and manual operation).

Muller resuscitator consists of a pneumatic valve feature designed to operate with medical oxygen. It is used intermittently or continuously for pulmonary re-expansion, with lower load imposed work, and increase the efficiency of gas exchange by improving volumes, lung capacity and breathing pattern, and reverse atelectasis.

However, studies show the paucity of data in the literature regarding the Muller Resuscitator in different forms and respiratory rehabilitation protocols. In addition, studies show lack of standardization of methods and resources used in respiratory therapy in patients with chest tube.

ELIGIBILITY:
Inclusion Criteria:

* Patients with old more 18 years untill 65 years
* Patients undergoing thoracic drainage
* That does not include in any exclusion criteria

Exclusion Criteria:

* Contraindications breathing equipment use positive pressure

  * Patient intolerance
  * Phobia
  * Hemodynamic instability
  * Use of vasopressiva therapy
  * Shock (systolic pressure <90 mmHg)
  * Face trauma
  * Nausea or vomiting
  * Acute myocardial infarction
  * Lobectomy
  * Lung cancer
  * Gastrointestinal surgery
  * Pleural fistula.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change Respiratory function | before the intervention (pre) and after drain removal the tube (pos) for 30 days
  Ventilometry was evaluated in two stages: 1) before the intervention, 2) on the day of drain removal or discharge. The spirometer application is according to implement stable and acceptable criteria. TOBIN The measures of lung volumes forão performed with the spirometer (FERRARIS MK8 Wright ®) coupled to a nozzle. The patient was instructed to breathe quietly in the apparatus for a minute to read the minute volume (VM). During this period, it is checked the number of breaths, i.e., respiratory rate (RR) for calculating the tidal volume (VT) given by VC = VM / FR (ml).

SECONDARY OUTCOMES:
Saturation Oxygen | 30 days
  Oxygen saturation was assessed in two stages: 1) before the first intervention of the day 2) after daily intervention protocol until hospital discharge or removal of the chest tube. Patients were evaluated with breathing in ambient air (without supplemental oxygen) after 10 minutes of the procedure. The researcher used a pulse oximeter portable.

OTHER OUTCOMES:
Pain | 30 days
  by visual analogue scale of pain (VAS) was used to determine the degree of soreness daily during the hospitalization period and pre chest drainage and after the intervention.
Hospitalization stay | 30 days
  the number of days in the hospital after chest drainage to discharge should be recorded for each patient. All patients were followed during hospitalization.
Time length chest drain | 30 days
  The length of the chest drain was checked until hospital discharge. The drain removal criterion was filed by the medical team of the hospital thoracic surgery. Debt drain in ml was collected by nursing professionals who were blinded study.
dyspnea | 30 days
  It was determined by the Borg scale, in two stages, before and after intervention in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula R Dos Anjos, mestranda, Principal Investigator — University of Campinas, Brazil
Locations (2):
- Brazil (2):
  - Hospital santa Casa de Passos, Passos, Minas Gerais
  - Hospital da Clínicas de campinas, Campinas, São Paulo

REFERENCES:
- [Background] Rahman NM, Chapman SJ, Davies RJ. Pleural effusion: a structured approach to care. Br Med Bull. 2005 Mar 14;72:31-47. doi: 10.1093/bmb/ldh040. Print 2004. PMID 15767562
- [Background] Hooper C, Lee YC, Maskell N; BTS Pleural Guideline Group. Investigation of a unilateral pleural effusion in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii4-17. doi: 10.1136/thx.2010.136978. No abstract available. PMID 20696692
- [Background] Porcel JM, Light RW. Diagnostic approach to pleural effusion in adults. Am Fam Physician. 2006 Apr 1;73(7):1211-20. PMID 16623208
- [Background] Woodrow P. Intrapleural chest drainage. Nurs Stand. 2013 Jun 5-11;27(40):49-56; quiz 58. doi: 10.7748/ns2013.06.27.40.49.e7373. PMID 23909181
- [Background] Kao JH, Kao HK, Chen YW, Yu WK, Pan SW, Wang JH, Lien TC, Ho LI, Kou YR. Impact and predictors of prolonged chest tube duration in mechanically ventilated patients with acquired pneumothorax. Respir Care. 2013 Dec;58(12):2093-100. doi: 10.4187/respcare.02273. Epub 2013 May 7. PMID 23651575
- [Background] Westerdahl E, Lindmark B, Almgren SO, Tenling A. Chest physiotherapy after coronary artery bypass graft surgery--a comparison of three different deep breathing techniques. J Rehabil Med. 2001 Mar;33(2):79-84. doi: 10.1080/165019701750098920. PMID 11474953
- [Background] Pasquina P, Tramer MR, Granier JM, Walder B. Respiratory physiotherapy to prevent pulmonary complications after abdominal surgery: a systematic review. Chest. 2006 Dec;130(6):1887-99. doi: 10.1378/chest.130.6.1887. PMID 17167013
- [Background] Hall JC, Tarala RA, Hall JL, Mander J. A multivariate analysis of the risk of pulmonary complications after laparotomy. Chest. 1991 Apr;99(4):923-7. doi: 10.1378/chest.99.4.923. PMID 2009796
- [Background] Muller AP, Olandoski M, Macedo R, Costantini C, Guarita-Souza LC. [Comparative study between intermittent (Muller Reanimator) and continuous positive airway pressure in the postoperative period of coronary artery bypass grafting]. Arq Bras Cardiol. 2006 Mar;86(3):232-9. doi: 10.1590/s0066-782x2006000300012. Epub 2006 Mar 30. Portuguese. PMID 16612452
- [Background] Ludwig C, Angenendt S, Martins R, Mayer V, Stoelben E. Intermittent positive-pressure breathing after lung surgery. Asian Cardiovasc Thorac Ann. 2011 Feb;19(1):10-3. doi: 10.1177/0218492310394664. PMID 21357311
- [Background] Catterall WA, Striessnig J. Receptor sites for Ca2+ channel antagonists. Trends Pharmacol Sci. 1992 Jun;13(6):256-62. doi: 10.1016/0165-6147(92)90079-l. PMID 1321525
- [Background] Holanda MA, Fortaleza SC, Alves-de-Almeida M, Winkeler GF, Reis RC, Felix JH, Lima JW, Pereira ED. Continuous positive airway pressure effects on regional lung aeration in patients with COPD: a high-resolution CT scan study. Chest. 2010 Aug;138(2):305-14. doi: 10.1378/chest.09-2850. Epub 2010 Apr 2. PMID 20363847